CLINICAL TRIAL: NCT03364075
Title: Genetic Variants Associated With the Occurrence of Localized Low Back Pain or Low Back Pain With Widespread Pain Symptoms, and Their Response to Treatment With Duloxetine or Propranolol
Brief Title: Genetic Variants Associated With Low Back Pain and Their Response to Treatment With Duloxetine or Propranolol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issue
Sponsor: Mark Ware (Other)
Responsible Party: Sponsor-Investigator, Mark Ware, BA, MBBS, MRCP, MSc, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MUHC15046
Record Dates: First submitted 2016-03-22; First posted 2017-12-06 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Duloxetine Hydrochloride; Propranolol; Genotype

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Duloxetine Treatment (Active Comparator): patients treated with Duloxetine
  Interventions: Drug: Duloxetine; Genetic: Genotype for SNPs associated to Serotonin and COMT; Drug: Placebo Treatment
- Propranolol Treatment (Active Comparator): patients treated with Propranolol
  Interventions: Drug: Propranolol; Genetic: Genotype for SNPs associated to Serotonin and COMT; Drug: Placebo Treatment
- Placebo Treatment (Placebo Comparator): patients treated with placebo
  Interventions: Drug: Duloxetine; Drug: Propranolol

INTERVENTIONS:
Drug: Duloxetine — 30 mg for seven days, then increased to 60 mg for seven days
  Other Names: Cymbalta
  Arms: Duloxetine Treatment; Placebo Treatment
Drug: Propranolol — 40 mg for seven days, then increase to 60 mg for seven days
  Other Names: TevaPropranolol
  Arms: Placebo Treatment; Propranolol Treatment
Genetic: Genotype for SNPs associated to Serotonin and COMT — DNA and RNA extraction from blood samples to identify genetic variants associated to pain pathways
  Arms: Duloxetine Treatment; Propranolol Treatment
Drug: Placebo Treatment — 1 capsule BID for two weeks
  Arms: Duloxetine Treatment; Propranolol Treatment

SUMMARY:
This study is a randomized, double-blind, placebo controlled, three period crossover clinical trial. The main purpose of this study is to determine if Chronic Low Back Pain patients presenting with either localized or widespread painful symptoms respond differently to treatment with Duloxetine or Propranolol, and if the effectiveness of treatment with these drugs can determined by the presence or absence of SNPs associated with the Serotonin receptor or Cathecol-O-MethylTransferase activity. Each treatment period will be of two weeks duration with a 1 week washout phase between treatment periods. Following a Latin square design, patients will be randomly assigned to one of six different treatment groups, starting their first treatment cycle with either Duloxetine, Propranolol or Placebo and rotating through the other treatments in the subsequent cycles. Effectiveness of treatment will be measured by means of Pain Index as the primary outcome measure, and secondary outcome measures will include Pressure Pain Threshold and the Pain Disability Index, Perceived Stress Scale, Symptom Checklist -90R and the Patient's Global Impression of Change questionnaires.

DETAILED DESCRIPTION:
Low back pain disorders are reported in 19-21% of the North American population, with the majority of them associating pain and physical impairment. Patients with this illness have an increased utilization of medical services, higher incidence of lost work days and long-term disability, representing a significant burden to the healthcare system and the economy.

Within the population of CLBP patients, two broad subgroups can easily be identified in the clinical setting: the patients who present with CLBP as their only pain symptom, and patients that present with CLBP and also associate widespread painful symptoms. The presence of widespread painful symptoms in the setting of low back pain has been recognized as a strong predictor of chronicity, apart from this, patients in this subgroup are more commonly middle aged females, report higher intensity of pain, more emotional problems and sleep disorders amongst others.

A recent publication by Slate et al has described genetic differences in patients with Temporal Mandibular Disorder (TMD) that present with either localized or widespread painful symptoms. This study established a link between Single Nucleotide Polymorphisms (SNPs) associated to the Serotonin Receptor and patients with localized TDM, and the presence of SNPs associated to the T cell receptor with patients with TMD and widespread symptoms. CLBP and TMD are two chronic pain conditions that are commonly present together. Given the connection between these two chronic pain disorders, it is highly likely that the genetic association findings from Slate et al could also be present in the CLPB population.

The main purpose of this study is to determine if CLBP patients presenting with either localized or widespread painful symptoms respond differently to treatment with Duloxetine, a Serotonin and Norepinephrine Reuptake Inhibitor (SNRI), and if the effectiveness of treatment with this drug can determined by the presence or absence of SNPs associated with the Serotonin receptor.

Another novel treatment alternative for patients with CLBP is Propranolol. This drug is a non-selective beta blocker that has also been shown to have analgesic effects on TMD. These effects though, are only present in patients carrying haplotypes associated with low activity of catechol-O-methyltransferase (COMT). The effect of beta blockers as analgesics has not yet been fully characterized, in animal models, catecholamine stimulation of beta 2 and beta 3 adrenoreceptors has shown to produce hyperalgesia and allodynia, on the other hand, in the clinical setting, the beta 1 selective blocker Esmolol has also been shown to have an analgesic effect in postoperative acute pain management. The inclusion of Propranolol as one of the treatment arms of this study will help elucidate Propranolol's possible role in chronic pain management; the expectation being that a more prominent analgesic effect will be found in patients displaying low activity COMT haplotypes.

Patients will be recruited from the Montreal General Hospital (MGH) Pain Centre and from the Quebec Pain Registry.

This study is a randomized, double-blind, placebo controlled, three period crossover clinical study. Each treatment period will be of two weeks duration with a 1 week washout phase between treatment periods. Following a Latin square design, patients will be randomly assigned to one of six different treatment groups, starting their first treatment cycle with either Duloxetine, Propranolol or Placebo and rotating through the other treatments in the subsequent cycles. The trial has a duration of 56 days total, and involves 6 clinic visits per participant, one at the beginning and at the end of each treatment cycle.

Randomization will be performed by a member of our research group that is not involved in the study using the online software (http//:www.randomization.com). The software's first generator will be used which randomizes each subject to a single treatment group by using the method of randomly permuted blocks. The randomization log will be provided to the pharmacy which will be in charge of dispensing the treatment.

All clinicians and researchers involved in the study data collection and experimental procedures will remain blinded to study group allocation for the duration of the study. Blinding will be maintained until the end for statistical analysis.

In case of serious adverse effects interfering with the patient safety, the blind responsible (pharmacy) will disclose the treatment to the MD of the MGH Pain Centre and that subject will be dropped out of the study.

ELIGIBILITY:
1. Male or Female patients aged 18 or above.
2. Chronic Low Back Pain as the primary painful condition. CLBP diagnose based on medical history and physical examination, with pain restricted to the low back (T6 or below), with or without radiation to the lower limbs but no neurologic signs defined as per the Quebec Task Force on Spinal Disorders Class 1 to 3. This pain must be persistent in the lower back ≥4 days/week for the past 6 months or longer.
3. Average pain score of ≥4 at the time of recruitment.
4. Women of childbearing potential must agree not to become pregnant during the time of the study and to use adequate contraception during this time. Adequate contraception will be defined as the use of highly effective or double barrier methods. When used consistently and correctly, "double barrier" methods of contraception (e.g. male condom with diaphragm, male condom with cervical cap) can be used as an effective alternative to the highly effective contraception methods such as combined oral contraceptives, injectables or intrauterine devices. Both options will be discussed during the informed consent process.
5. Stable drug regimen for 1 month prior to entering the study and throughout the study. Patients will not be taken off their current pain medication to participate in the study, but they will be asked to keep a stable regimen (not change any doses, add or remove other medication) during the study.
6. Ability to follow study protocol (cognitive and situational).
7. Ability to write and speak in English and/or French.
8. Agrees to provide signed and dated informed consent form and biobanking consent form.
9. Willing to comply with all study procedures, including the biobanking aspect of the project and to be available for the duration of the study.

Exclusion Criteria:

1. Uncontrolled medical or psychiatric conditions.
2. History of major depressive disorder, psychotic disorder or schizophrenia, and/or manic episodes within the past year.
3. Pregnancy and/or breast-feeding. Patients who are unsure of their status will also be excluded from participating
4. Pain due to cancer.
5. Disability compensation or litigation.
6. Neurologic signs of lumbosacral radiculopathy within the past 6 months: lower extremity muscle weakness/sensory loss in a dermatomal distribution, abnormal deep tendon reflexes.
7. Radiographic and/or electrophysiology evidence of radicular compression in the past 6 months.
8. Clinical signs of lumbar stenosis within the past 6 months: numbness, weakness, and/or discomfort radiating from the spine down to the buttocks and legs while walking or in prolonged standing and relieved with sitting or lying.
9. Clinical signs of back pain that requires an urgent/alternative intervention: new onset bowel/bladder incontinence, saddle anaesthesia, foot drop, unexplained weight loss, fever.
10. Radiographic evidence of spinal stenosis, high-grade spondylolisthesis (grade 3 or 4), acute spinal fracture, tumour, abscess or acute pathology in the low back/abdominal area in the past 6 months.
11. Low back surgery (lumbosacral spine) within the past 12 months, or history of more than 1 low back surgery.
12. Minimally invasive procedures aimed to reduce pain in the lumbosacral area within the past month (Medial Branch Blocks/Ablations, Epidural Steroid Injections, Trigger point injections, Sacroiliac Joint Injections, Greater Trochanteric/Acetabulofemoral Joint Injections).
13. Known hypersensitivity to Beta Blockers or SNRIs.
14. Currently taking SNRIs, Beta Blockers, Opioids at a daily dose superior to 30mg of Morphine Oral Equivalent, Tricyclic Antidepressants, Methylene Blue, Linezolid, Monoamine Oxidase Inhibitors (such as Selegiline, Isoniazid, Procarbazine), Thioridazine, CYP1A2 inhibitors (Fluvoxamine, Verapamil, Cimetidine, Fluoroquinolone antibiotics such as Ciprofloxacin).
15. Active alcoholism within the past 6 months.
16. Psychoactive recreational drug abuse within the past 6 months including MDMA, Ketamine, hallucinogens such as LSD and/or sympathomimetics such as Cocaine.
17. Patients with asthma, cardiac arrhythmias such as Wolff-Parkinson-White syndrome, coronary artery disease, congestive heart failure, renal failure or dialysis, liver insufficiency, diabetes mellitus, hyperthyroidism.
18. Heart rate less than 60 bpm or systolic/diastolic blood pressure less than 105/60 mmHg during the initial visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
pain index | Difference between the average pain index on the first three days of treatment compared to the last three days of the 14 day treatment cycle
  Average pain intensity multiplied by percentage of time in pain in the waking day.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ware, MBBS MRCP, Principal Investigator — Director of Clinical Research Alan Edwards Pain Management Unit
Locations (1):
- Centre for Innovative Medicine - McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim KL, Jacobs P, Klarenbach S. A population-based analysis of healthcare utilization of persons with back disorders: results from the Canadian Community Health Survey 2000-2001. Spine (Phila Pa 1976). 2006 Jan 15;31(2):212-8. doi: 10.1097/01.brs.0000194773.10461.9f. PMID 16418643
- [Background] Von Korff M, Crane P, Lane M, Miglioretti DL, Simon G, Saunders K, Stang P, Brandenburg N, Kessler R. Chronic spinal pain and physical-mental comorbidity in the United States: results from the national comorbidity survey replication. Pain. 2005 Feb;113(3):331-339. doi: 10.1016/j.pain.2004.11.010. PMID 15661441
- [Background] Coyte PC, Asche CV, Croxford R, Chan B. The economic cost of musculoskeletal disorders in Canada. Arthritis Care Res. 1998 Oct;11(5):315-25. doi: 10.1002/art.1790110503. PMID 9830876
- [Background] Koes BW, van Tulder M, Lin CW, Macedo LG, McAuley J, Maher C. An updated overview of clinical guidelines for the management of non-specific low back pain in primary care. Eur Spine J. 2010 Dec;19(12):2075-94. doi: 10.1007/s00586-010-1502-y. Epub 2010 Jul 3. PMID 20602122
- [Background] Fairbank J, Gwilym SE, France JC, Daffner SD, Dettori J, Hermsmeyer J, Andersson G. The role of classification of chronic low back pain. Spine (Phila Pa 1976). 2011 Oct 1;36(21 Suppl):S19-42. doi: 10.1097/BRS.0b013e31822ef72c. PMID 21952188
- [Background] Thomas E, Silman AJ, Croft PR, Papageorgiou AC, Jayson MI, Macfarlane GJ. Predicting who develops chronic low back pain in primary care: a prospective study. BMJ. 1999 Jun 19;318(7199):1662-7. doi: 10.1136/bmj.318.7199.1662. PMID 10373170
- [Background] Natvig B, Bruusgaard D, Eriksen W. Localized low back pain and low back pain as part of widespread musculoskeletal pain: two different disorders? A cross-sectional population study. J Rehabil Med. 2001 Jan;33(1):21-5. doi: 10.1080/165019701300006498. PMID 11480465
- [Background] Slade GD, Smith SB, Zaykin DV, Tchivileva IE, Gibson DG, Yuryev A, Mazo I, Bair E, Fillingim R, Ohrbach R, Greenspan J, Maixner W, Diatchenko L. Facial pain with localized and widespread manifestations: separate pathways of vulnerability. Pain. 2013 Nov;154(11):2335-2343. doi: 10.1016/j.pain.2013.07.009. Epub 2013 Jul 16. PMID 23867732
- [Background] Wiesinger B, Malker H, Englund E, Wanman A. Back pain in relation to musculoskeletal disorders in the jaw-face: a matched case-control study. Pain. 2007 Oct;131(3):311-319. doi: 10.1016/j.pain.2007.03.018. Epub 2007 Apr 24. PMID 17459585
- [Background] Millan MJ. Descending control of pain. Prog Neurobiol. 2002 Apr;66(6):355-474. doi: 10.1016/s0301-0082(02)00009-6. PMID 12034378
- [Background] Tchivileva IE, Lim PF, Smith SB, Slade GD, Diatchenko L, McLean SA, Maixner W. Effect of catechol-O-methyltransferase polymorphism on response to propranolol therapy in chronic musculoskeletal pain: a randomized, double-blind, placebo-controlled, crossover pilot study. Pharmacogenet Genomics. 2010 Apr;20(4):239-48. doi: 10.1097/FPC.0b013e328337f9ab. PMID 20216107